CLINICAL TRIAL: NCT02379559
Title: An Exercise Intervention on Metabolic Syndrome and Prostate Cancer Risk Among Black Men
Brief Title: Exercise Intervention Metabolic Syndrome Prostate Cancer Black Men
Acronym: STRONG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Georgetown_University_MC1
Record Dates: First submitted 2014-09-23; First posted 2015-03-05 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2014-09

CONDITIONS: Physical Activity; Metabolic Syndrome; Prostate Cancer
Keywords: prostate cancer; African-American; Metabolic Syndrome; Exercise; Men's Health
MeSH Terms: conditions — Motor Activity; Metabolic Syndrome; Prostatic Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise Group (Experimental): Eligible participants randomized into the intervention group will receive a mix of supervised moderate-intensity aerobic and light weight-resistance exercises.
  Interventions: Behavioral: Exercise
- Attention Control Group (Active Comparator): Eligible participants randomized in the attention control group will be asked to maintain their current daily activities and exercise habits for 6-months.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Exercise — For the first 12-weeks, participants will come to our community based research office for up to 50 min/session, 3-days/week of supervised exercise. Exercise duration will increase from 75 min/wk at week 1 to 150 min/wk by week 4. Thereafter, men will maintain 150 min/wk of moderate-intensity physical activity.
  Arms: Exercise Group
Behavioral: Attention Control — We will provide weekly healthy lifestyle tips via text messages, and will include tips such as managing stressors in life and getting better sleep.
  Arms: Attention Control Group

SUMMARY:
The main purpose of this study is to examine the feasibility of an exercise intervention on metabolic syndrome (MetS) components and biomarkers related to prostate cancer in Black men with MetS who are at increased risk of prostate cancer.

DETAILED DESCRIPTION:
The specific aim for the proposed study is to examine the feasibility and impact of a 6-month two-arm randomized controlled trial (RCT) on MetS components and biomarkers related to prostate cancer in Black men with MetS. Due to the striking racial disparities of prostate cancer, this proposal will focus on the impact of an aerobic and resistance exercise intervention on MetS and biomarkers related to prostate cancer in Black men. Specifically, our proposed clinical trial compares an aerobic and resistance exercise intervention to an attention control group among Black men.

ELIGIBILITY:
Inclusion Criteria:

1. African-American and/or Black men;
2. between the ages of 40-70 years;
3. waist circumference >40 inches (102 cm);
4. with at least two of the following: elevated BP (≥ 130/85 mmHg);
5. elevated fasting glucose (≥ 100 mg/dL), reduced HDL cholesterol (<50 mg/dL), or elevated triglycerides (≥ 150 mg/dL);
6. sedentary defined as <60 minutes of recreation or work requiring modest PA/week;
7. be able to speak and read English;
8. able to provide meaningful consent (i.e., men with severe cognitive impairment will be excluded);
9. have no physical limitations that prevent from exercising;
10. and have access to a television and DVD player.

Exclusion Criteria:

1. history of cancer except nonmelanoma skin cancer;
2. current enrollment in another clinical trial or weight loss program;
3. inability to commit to the intervention schedule. Prior to randomization, participants will be required to have a signed authorization and medical clearance from their personal physician or our nurse practitioner.

Ages: 40 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-07; Primary Completion 2017-02-16 (Actual); Study Completion 2017-02-16 (Actual)

PRIMARY OUTCOMES:
Waist circumference | 6-months
  Waist circumference will be measured at baseline, 3- and 6-months of the intervention

SECONDARY OUTCOMES:
Dietary behaviors questionnaire | 6-months
  Block 2005 Food Frequency Questionnaires (FFQ) at baseline, 3- and 6-months of the intervention
Cardiovascular fitness test | 6-months
  Bruce treadmill protocol will be used to determine VO2max at baseline, 3- and 6-months of the intervention.
Fasting glucose levels test | 6-months
  Fasting blood sample via finger sticks will be administered by a phlebotomist to measure fasting glucose levels at baseline, 3- and 6-months of the intervention.
Lipid level test | 6-months
  Fasting blood sample via finger sticks will be administered by a phlebotomist to measure lipid levels at baseline, 3- and 6-months of the intervention.
Quality of life questionnaire (SF-36) | 6-months
  Short Form 36 Health Survey (SF-36) will be administered at baseline, 3- and 6-months of the intervention.
Body Mass Index (BMI) | 6-months
  Weight (lbs) and height (inches) will be measured to calculate BMI at baseline, 3- and 6-months of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Office of Minority Health and Health Disparities Research, Washington D.C., District of Columbia, United States